CLINICAL TRIAL: NCT00517218
Title: A Randomized Phase 3 Study of Fludarabine and Rituximab With or Without Genasense® (Oblimersen Sodium) in Previously Untreated Subjects With Chronic Lymphocytic Leukemia
Brief Title: This Study is Being Performed to Evaluate the Effect of Genasense on the Efficacy and the Safety of Rituximab/Fludarabine Combination Treatment in Previously Untreated Subjects With Chronic Lymphocyctic Leukemia(CLL)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL305
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2007-08

CONDITIONS: Lymphocytic Leukemia
Keywords: Evaluate the Effect of Genasense on the Efficacy/Safety of Rituximab/Fludarabine Treatment in Untreated Subjects With Chronic Lymphocyctic Leukemia
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — oblimersen

INTERVENTIONS:
Drug: Genasense® (, oblimersen sodium G3139)

SUMMARY:
To compare the efficacy and safety of combination treatment with Genasense, fludarabine, and rituximab versus combination treatment with fludarabine and rituximab in previously untreated subjects with CLL.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated subjects with intermediate-or high-risk CLL(modified Rai Stages I-IV)
* Measurable disease as primarily established by the National Cancer Institute-sponsored Working Group(NCI-WG) Guidelines for the diagnosis of CLL
* Requiring therapy for active disease, as primarily defined by the NCI-WG Guidelines
* Eastern Cooperative Oncology Group Performance Status < 2
* Adequate organ function determined , 14 days prior to the first dose of study medication

Exclusion Criteria:

* Absolute Lymphocyte count > 100,000/uL
* Prior chemotherapy or other therapy for CLL, including allogeneic transplant
* Less than 3 weeks from any prior major surgery at the time of informed consent
* Failure to recover from any serious adverse effect of surgery
* History of autoimmune hemolytic anemia or autoimmune thrombocytopenia
* Active serious infection requiring systemic anti-infective therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Study Completion 2009-06